CLINICAL TRIAL: NCT00430872
Title: Validation of the M.D. Anderson Symptom Inventory-Spine Tumor Module
Brief Title: Development of the MDASI-Spine Tumor Module
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0809
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Spinal Cord Tumor
Keywords: Spinal Cord Tumor; Intramedullary Spinal Cord Tumor; Extramedullary Spinal Cord Tumor; Symptoms; Survey
MeSH Terms: conditions — Spinal Cord Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MDASI-Spine Tumor Module Survey: M. D. Anderson Symptom Inventory-Spine (survey) of patients with a tumor on the spine or spinal cord.
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — Survey about the severity of certain symptoms lasting 10-15 minutes.
  Other Names: MDASI-Spine

SUMMARY:
The goal of this research study is to learn the severity of certain symptoms in patients with tumors of the spine or spinal cord. Researchers also want to learn if the M. D. Anderson Symptom Inventory-Spine is a good way to rate these symptoms.

Primary Objective:

1. To evaluate the psychometric properties of the MDASI-Spine in patients with tumors involving the spine or spinal cord.

Secondary Objective:

1. To describe the severity of commonly occurring symptoms experienced by persons with spine tumors.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will complete the M. D. Anderson Symptom Inventory-Spine Tumor Module survey. This survey will ask you to rate the severity of certain symptoms you may have had in the last 24 hours on a scale of 0 (not present) to 10 (the most severe you can imagine). You will also be asked to rate how your symptoms get in the way of your daily activities using the same 0 to 10 scale. This survey should take about 10-15 minutes to complete.

Information regarding your clinical history (tumor type, location, treatment, and other medications) and demographic information (age, gender, ethnicity, religion, educational level, and marital status) will also be collected. This information will be used to evaluation whether there is an association between symptom severity and these factors.

Once you have completed the survey, your participation on this study will be over.

This is an investigational study. Up to 128 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of a tumor involving the spinal cord (intramedullary or extramedullary)
2. Age > or = to 18 years of age
3. Ability to speak and read English. Non-English speaking subjects will be included in future studies, once the final instrument has been developed.

Exclusion Criteria:

1. Patients < 18 years of age
2. Evidence of gross cognitive dysfunction limiting memory or ability to complete a self-report questionnaire as determined by evaluation of physician or mid-level provider.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a tumor on the spine or spinal cord.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Overall MDASI Score | 18 Months

SECONDARY OUTCOMES:
Proportion of Patients Reporting Symptom Severity >4 on 0-10 Scale | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Terri S. Armstrong, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org